CLINICAL TRIAL: NCT00140530
Title: A Randomized Trial of a Nonpolymer-Based Rapamycin-Eluting Stent Versus a Polymer-Based Paclitaxel-Eluting Stent for the Prevention of Restenosis (ISAR-TEST-1)
Brief Title: Nonpolymer- and Polymer-Based Drug-Eluting Stents for Restenosis (ISAR-TEST-1)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Bayerische Forschungsstiftung Muenchen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02103; AZ 504/02
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Due to randomisation patients got a Paclitaxel-eluting stent
  Interventions: Device: Paclitaxel-eluting stent (Taxus)
- 2 (Experimental): Due to randomization patients got a Rapamycin-eluting stent.
  Interventions: Device: Rapamycin-eluting stent

INTERVENTIONS:
Device: Paclitaxel-eluting stent (Taxus) — patients has been implanted the Paclitaxel-eluting stent.
  Other Names: Taxus
  Arms: 1
Device: Rapamycin-eluting stent — patients has been implanted the Rapamycin-eluting stent.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of nonpolymer-based rapamycin-eluting stent compared to standard polymer-based paclitaxel-eluting stent to reduce reblockage of coronary arteries.

DETAILED DESCRIPTION:
Drug-eluting stents represent a major advance in the treatment of restenosis. They have dramatically reduced the need of repeat revascularization procedures, and, thanks to the excellent results obtained in various patient subsets, these devices are now used in almost 90% of the stent implantation procedures performed in US hospitals. Along with the increasing number of patients receiving drug-eluting stents and availability of long-term follow-up data, concern has arisen regarding the safety of these devices. At the core of this concern is the potential for increased inflammatory and thrombogenic responses and their life-threatening consequences associated with the polymers employed for the delivery of antirestenotic agents. A growing interest has been shown on polymer-free stents with a microporous surface as an alternative to stents employing polymeric coating for local drug delivery. Recently, we developed a mobile system which enables coating in the catheterization laboratory of polymeric free stents with different drug doses or combinations. Using a porcine coronary model of restenosis, we found that coating with rapamycin of a polymer-free microporous stent is feasible and effectively reduces neointimal proliferation. More recently, in a clinical study in which the efficacy of several doses of rapamycin was assessed, we showed that non-polymer coating with rapamycin is safe and leads to a dose-dependent reduction in restenosis. While the advantage deriving from the lack of polymeric cover in on-site coated rapamycin-eluting stents is readily understandable, their relative efficacy as compared with commercially available polymer-based drug-eluting stents has yet to be evaluated.

Comparison:

Polymer-free microporous stents coated with rapamycin versus standard polymer-based, paclitaxel-eluting stents

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Stable or unstable angina or a positive stress test
* "de novo" coronary artery lesions
* Written informed consent

Exclusion Criteria:

* Myocardial infarction within 48 h. before enrollment
* Target lesion located in left main trunk
* Contraindication or known allergy to aspirin, heparin, thienopyridines, rapamycin, paclitaxel or stainless steel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2004-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
In-stent late luminal loss | 6 months

SECONDARY OUTCOMES:
Angiographic restenosis at follow-up angiography | 6 months
Need for target lesion revascularization due restenosis at 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Hausleiter J, Kastrati A, Wessely R, Dibra A, Mehilli J, Schratzenstaller T, Graf I, Renke-Gluszko M, Behnisch B, Dirschinger J, Wintermantel E, Schomig A; investigators of the individualizable durg-eluting Stent System to Abrogate Restenosis Project. Prevention of restenosis by a novel drug-eluting stent system with a dose-adjustable, polymer-free, on-site stent coating. Eur Heart J. 2005 Aug;26(15):1475-81. doi: 10.1093/eurheartj/ehi405. Epub 2005 Jun 23. PMID 15975990
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Virmani R, Liistro F, Stankovic G, Di Mario C, Montorfano M, Farb A, Kolodgie FD, Colombo A. Mechanism of late in-stent restenosis after implantation of a paclitaxel derivate-eluting polymer stent system in humans. Circulation. 2002 Nov 19;106(21):2649-51. doi: 10.1161/01.cir.0000041632.02514.14. PMID 12438288
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Result] Mehilli J, Kastrati A, Wessely R, Dibra A, Hausleiter J, Jaschke B, Dirschinger J, Schomig A; Intracoronary Stenting and Angiographic Restenosis--Test Equivalence Between 2 Drug-Eluting Stents (ISAR-TEST) Trial Investigators. Randomized trial of a nonpolymer-based rapamycin-eluting stent versus a polymer-based paclitaxel-eluting stent for the reduction of late lumen loss. Circulation. 2006 Jan 17;113(2):273-9. doi: 10.1161/CIRCULATIONAHA.105.575977. Epub 2006 Jan 3. PMID 16391155
- [Derived] King L, Byrne RA, Mehilli J, Schomig A, Kastrati A, Pache J. Five-year clinical outcomes of a polymer-free sirolimus-eluting stent versus a permanent polymer paclitaxel-eluting stent: final results of the intracoronary stenting and angiographic restenosis - test equivalence between two drug-eluting stents (ISAR-TEST) trial. Catheter Cardiovasc Interv. 2013 Jan 1;81(1):E23-8. doi: 10.1002/ccd.24375. Epub 2012 May 4. PMID 22431239